CLINICAL TRIAL: NCT06448923
Title: Effects of an Acute 1-month Cannabidiol Treatment on Pain and Inflammation After a Long Bone Fracture: a Triple-blind Randomized, Placebo Controlled Clinical Trial
Brief Title: Cannabidiol After Multi-Trauma for Pain and Opioid Therapy
Acronym: CAM-POT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Louis De Beaumont, Principal Investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-2105
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Fracture
Keywords: Cannabidiol; Trauma; Pain; Inflammation; Fracture; Orthopaedic
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries; Pain; Inflammation | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low CBD dose (Experimental): Participants will receive 25 mg orally twice daily during a meal for a month
  Interventions: Drug: Cannabidiol
- Moderate CBD dose (Experimental): Participants will receive 50 mg orally twice daily during a meal for a month
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Participants will receive matching placebo orally twice daily during a meal for a month
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — 25 mg of CBD tablets twice daily
  Arms: Low CBD dose
Drug: Cannabidiol — 50 mg of CBD tablets twice daily
  Arms: Moderate CBD dose
Drug: Placebo — Matching placebo tablets twice daily
  Arms: Placebo

SUMMARY:
The aim of this project is to investigate the therapeutic potential and safety of acute Cannabidiol (CBD) treatment on longitudinal pain symptoms, and to assess potential interactions with pain mediators including opioids and sex on CBD treatment response. To this end, this research protocol proposes a comprehensive translational approach including a placebo-controlled randomized clinical trial comparing two daily doses of CBD treatment administered for one month on pain relief. This study will also compare intervention conditions on inflammation markers, participant quality of life, sleep quality, depression, anxiety, cognition and orthopaedic function.

DETAILED DESCRIPTION:
The level of pain in the acute phase after injury is a predictor of the development of chronic pain. Chronic pain is defined as pain that persists for more than 3 months post-accident and impairs functional recovery. Mechanistically, it has been shown that acute nonspecific inflammation triggered after peripheral injury results in the continuous release of proinflammatory cytokines that weaken the blood-brain barrier, facilitating the entry of toxins that can invade the central nervous system (CNS). The resulting sustained inflammation of the CNS plays an important role in establishing the maladaptive plasticity process underlying pain chronification. Cannabidiol (CBD), a component of cannabis devoid of addictive or psychotropic effects, stands out as a potential therapeutic agent given its analgesic and anti-inflammatory properties as well as its potential to enhance the biomechanical properties of bone healing. Given the excellent safety profile of CBD and its inhibitory effects on microglial activity, the primary mechanism of neuroinflammation and pain, CBD has the potential to promote acute pain relief while reducing reliance on addictive opioid treatments, hence facilitating recovery in trauma patients.

This study is a randomized, placebo controlled, human pilot clinical trial evaluating the effects of two doses (low and moderate) of CBD vs. placebo on pain after orthopaedic trauma.

Risks of adverse effects are considered low given the demonstrated excellent safety profile of CBD. CBD was also shown to accentuate opioid analgesic effects, thus reducing required opioid doses for patient comfort. The most likely adverse events associated with CBD in adult patients include somnolence, fatigue, drowsiness and decreased appetite. Access to on-duty emergency physicians at the recruiting site will be provided during the entire treatment duration.

A 30% relative pain intensity reduction on the VAS (expected response of 50% or more in the CBD group and expected 20% in the placebo group) has been used extensively to reflect clinically significant pain relief in clinical trials. Based on a Fisher's exact test, a sample size of 225 participants (3 groups of 75) will be required to reach a power of 80% to detect a statistically significant difference in the proportion of patients who reaches 30% pain reduction between the CBD groups and placebo at 1-month post-injury, assuming a dropout rate of 20% and a significance level of 5%. These parameters are taken from a successful randomised, placebo-controlled clinical trial using Sativex© in treating 125 neuropathic pain patients. Moreover, considering that the placebo group may ingest more opiates and that the anticipated inter-group effect at one month may be reduced to 20%, a total sample size of 225 subjects could be required to achieve 80% power, assuming a drop-out rate of 20% and a significance level of 5%.

Our group has ensured the feasibility of conducting such a pilot clinical trial in multi-trauma patients with the recruitment of 110 patients in less than 18 months to take part in a 10-session, outpatient treatment trial. A partnership with Canadian company EmpowerPharm will enable the use of pharmaceutical-grade synthetic CBD samples and identical placebos. The pharmacokinetic profile of the CBD product has been established.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a long bone fracture of the lower limb (tibia, fibula, femur, metatarsals, and phalanges) or the upper limb (humerus, radius, ulna, metacarpals, and phalanges) treated to Sacre-Coeur Hospital in Montreal (HSCM) within one week of the accident
* Participants is between 18 and 70 years of age
* Patients with or without surgical procedures

Exclusion Criteria:

* Moderate/severe traumatic brain injury (TBI)
* Diagnosis of any of the following mental disorders as defined by the DSM-5: schizophrenia, intellectual disability, bipolar disorder, major depression, a diagnosed and untreated sleep disorders
* History of alcohol or opioid misuse/abuse, as defined by the DSM-5
* Evidence of severe renal (stage 4 or 5) or hepatic impairment (Child B or C)
* Pregnant or lactating women, women of childbearing potential who are not using medically accepted forms of contraception (e.g., condoms, oral contraceptive or intrauterine device), or women who are actively planning on becoming pregnant
* History of adverse reactions to cannabis
* Patients taking warfarin, sildenafil, valproate or under opioids treatment prior to the injury
* Patients experiencing on average mild-to-absent pain in the last 24h preceding recruitment (as per a score <30 on a 0-100mm Visual Analogue Scale (VAS))
* Transport business drivers and heavy machinery operators
* A diagnosis of chronic pain, bone pathology (e.g., osteoporosis) or chronic inflammatory disease (e.g., rheumatoid arthritis, arthritis, psoriasis)
* Not having French or English as a spoken language
* A weighted MoCA score of less than 24
* Regular cannabis use more than 5 times a week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline on Pain Intensity Rating on a Visual Analog Scale (VAS) at Week 4 | Baseline and 4 weeks
  VAS pain intensity will be collected at baseline (before the start of treatment), twice a week during treatment, 24 hours after the end of treatment and at the 3-month follow-up. The VAS is a 100 mm line with anchor words ranging from "no pain" to "worst pain imaginable". Participants will be asked to place an intersecting mark along the line to indicate their pain intensity at the specific time of the test.

SECONDARY OUTCOMES:
Response Rate - 50 Percent or Greater Reduction in Pain Intensity on a Visual Analog Scale (VAS) | 4 weeks
  The response rate was defined as the number of participants with a 50 percent or greater reduction in VAS pain score from baseline to end of treatment. The VAS is a 100 mm line with anchor words ranging from "no pain" to "worst pain imaginable".
Change in Pain Rating on the Brief Pain Inventory Short Form (BPI-sf) Between Interventions | 4 weeks and 3 months
  The Brief Pain Inventory short form (BPI-sf) is a 9-item self-reported questionnaire assessing for the presence, intensity, and location(s) of pain, as well as perceived efficacy of pain relief treatment, and pain interference with activities of daily living. Item scores range from 0-10. The lower the score, the better the subject's pain.
Change in Blood Level Inflammation Over Time and Between Interventions | Baseline, 4 weeks and 3 months
  Blood levels of pro-inflammatory cytokines including interleukins (IL-6, IL-10) and tumor necrosis factor-alpha (TNF-α) will be collected and quantified.
Opioid Usage Monitoring | Ongoing from baseline to 3 months
  Opioid usage will be collected from daily medication diary for the first month and from number of prescription refills for months 2 and 3.
Change in the Orthopaedic Function Using The Short Musculoskeletal Function Assessment (SMFA) Questionnaire Between Interventions | 4 weeks and 3 months
  The SMFA consists of 34 questions covering the assessment of the patients function and 12 questions related to how bothered patients are by their symptoms. All categories are scored together, totaling between 0-100 percent. The lower the score, the better the subject's function.
Change in Quality of Life Using the Short Form (36) Health Survey Between Interventions | 4 weeks and 3 months
  The SF-36 is a 36-item self-report questionnaire for measuring quality of life across 9 domains. Scores range from 0-100, the lower the score, the worse is the subject's quality of life.
Change in Sleep Quality Using the Pittsburgh Sleep Quality Index (PSQI) Between Interventions | 4 weeks and 3 months
  A self-report questionnaire that assesses sleep quality and quantity during the past 4 weeks. The PSQI contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Change in Depression Symptoms Assessment Using the Beck's Depression Inventory-II Between Interventions | Baseline, 4 weeks and 3 months
  A 21-item multiple-choice self-report questionnaire for measuring depression symptoms. Scores range from 0 to 63, with higher scores representing more severe symptoms of depression.
Change in Anxiety Symptoms Assessment Using the Beck's Anxiety Inventory Between Interventions | Baseline, 4 weeks and 3 months
  A 21-question multiple-choice self-report inventory used for measuring the severity of anxiety symptoms. Score range from 0 to 63. Higher scores indicate more severe anxiety symptoms.
Change in Speed of Information Processing using Symbol Search from the WAIS-IV Battery Between Intervention | Baseline, 4 weeks and 3 months
  A neuropsychological test highly sensitive to both mild traumatic brain injury (mTBI) and pain and which do not require the use of injured limbs will be administered. Symbol Search from the WAIS-IV Battery, a tasks assessing speed of information processing, will be administered. Scaled Score range from 0 to 19. Higher scores indicate better processing speed.
Change in Attention using Elevator counting with distraction from the Test of Everyday Attention Battery Between Intervention | Baseline, 4 weeks and 3 months
  A neuropsychological test highly sensitive to both mild traumatic brain injury (mTBI) and pain and which do not require the use of injured limbs will be administered. Elevator counting with distraction from the Test of Everyday Attention Battery, a tasks assessing attention, will be administered. Scaled Score range from 0 to 19. Higher scores indicate better attention.
Change in Attention using Elevator counting from the Test of Everyday Attention Battery Between Intervention | Baseline, 4 weeks and 3 months
  A neuropsychological test highly sensitive to both mild traumatic brain injury (mTBI) and pain and which do not require the use of injured limbs will be administered. Elevator counting from the Test of Everyday Attention Battery, a tasks assessing attention, will be administered. Scaled Score range from 0 to 19. Higher scores indicate better attention.
Change in Memory using the California Verbal Learning Test Between Interventions | Baseline, 4 weeks and 3 months
  A neuropsychological test highly sensitive to both mild traumatic brain injury (mTBI) and pain and which do not require the use of injured limbs will be administered. The California Verbal Learning Test, a tasks assessing memory, will be administered. Standard Score range from -5 to 5. Higher scores indicate better memory.
Change in Memory using Digit Span from the WAIS-IV Battery Between Intervention | Baseline, 4 weeks and 3 months
  A neuropsychological test highly sensitive to both mild traumatic brain injury (mTBI) and pain and which do not require the use of injured limbs will be administered. Digit Span from the WAIS-IV Battery, a tasks assessing memory, will be administered. Scaled Score range from 0 to 19. Higher scores indicate better memory.
Change in Executive Fonction using the D-KEFS Color-Word Between Interventions | Baseline, 4 weeks and 3 months
  A neuropsychological test highly sensitive to both mild traumatic brain injury (mTBI) and pain and which do not require the use of injured limbs will be administered. The D-KEFS Color-Word, a tasks assessing executive function, will be administered. Scaled Score range from 1 to 19. Higher scores indicate better executive function.
Change in Executive Function using the D-KEFS Verbal Fluency Between Interventions | Baseline, 4 weeks and 3 months
  A neuropsychological test highly sensitive to both mild traumatic brain injury (mTBI) and pain and which do not require the use of injured limbs will be administered. The D-KEFS Verbal Fluency, a tasks assessing executive function, will be administered. Scaled Score range from 1 to 19. Higher scores indicate better executive function.

OTHER OUTCOMES:
Pain catastrophization using the Pain Catastrophizing Scale | Baseline
  The Pain Catastrophizing Scale is a 15-item self-report questionnaire assessed with Likert Scales. The overall score has a range of 0-52, with higher scores representing more severe symptoms.
Change in mTBI symptoms resolution using the Rivermead Post-Concussion Questionnaire (RPQ) | Baseline, 4 weeks and 3 months
  Only for participants diagnosed with mTBI related to the injury. The RPQ has a total possible score of 0-52, with higher scores indicative of worse outcomes.
Treatment Expectation using the Treatment Expectation Questionnaire (TEX-Q-F) | Baseline
  The Treatment Expectation Questionnaire is a 15-item questionnaire assessing the level of expectation towards treatment. The scale of the items ranges from 0 to 10. Higher scores indicate higher expectations.
Symptoms of Post-Traumatic Stress Disorder using the PTSD Checklist for DSM-5 (PCL-5) questionnaire | Baseline and 4 weeks
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure of the Diagnostic and Statistical Manual (DSM-5) symptoms of PTSD. Scores range from 0 to 80, with higher scores representing more severe symptoms of PTSD.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Sacré-Coeur de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Brazeau D, Deshaies AA, Williamson D, Bernard F, Arbour C, Pinard AM, Rouleau D, De Beaumont L. Impact of an acute 1-month cannabidiol treatment on pain and inflammation after a long bone fracture: a triple-blind randomised, placebo-controlled, clinical trial protocol. BMJ Open. 2025 Feb 20;15(2):e092919. doi: 10.1136/bmjopen-2024-092919. PMID 39979051